CLINICAL TRIAL: NCT05711459
Title: A Prospective and Multicenter Cohort Study of Bicyclol in the Treatment of Antineoplastic Drug-induced Liver Injury.
Brief Title: Bicyclol in the Treatment of Antineoplastic Drug-induced Liver Injury.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDILI
Record Dates: First submitted 2022-11-13; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-12

CONDITIONS: Drug-Induced Acute Liver Injury
Keywords: Prospective Study; Multicenter Trials; Bicyclol Tablet; Antineoplastic Drug-induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — bicyclol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Injury Group (Experimental): The patients have liver injuries caused by antitumor drugs.
  Interventions: Drug: Bicyclol tablets

INTERVENTIONS:
Drug: Bicyclol tablets — Take Bicyclol tablets for the treatment of liver injury.

SUMMARY:
The clinical trial is designed to evaluate the efficacy of bicyclol for patients with antineoplastic drug-induced liver injury and investigate factors effecting the therapeutic outcome.

DETAILED DESCRIPTION:
This study prospectively studied the treatment of acute drug-induced liver injury related to anti-tumor with bicyclol tablets, to provide medical evidence in clinical practice of bicyclol treating acute drug-induced liver injury. The main purpose of this study is to evaluate the clinical efficacy and outcome of bicyclol tablets in the treatment of drug-induced liver injury and analyze the bicyclol tablet's therapeutic effects in different groups including conventional chemotherapy drugs, targeted drugs, and immunosuppressants. The secondary purpose of this study is to analyze the factors influencing the prognosis and outcome of bicyclol tablets in the treatment of acute DILI.

ELIGIBILITY:
Inclusion Criteria:

1. The acute liver injury caused by anti-tumor drugs
2. The RUCAM assessment scale ≥6
3. The liver injury must in the acute phase
4. Must be treated with bicyclol tablets
5. Must sign informed consent -

Exclusion Criteria:

1. This acute liver injury caused by non-anti-tumor drugs
2. Pregnant women
3. Lactating women
4. Childbearing age women are plan to conceive

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5405 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The changes in ALT level from baseline after 4 weeks treatment of bicyclol | 4 weeks
  Excellence: clinical symptoms and signs disappeared, serum ALT returned to normal; Improvement: clinical symptoms disappeared (improved), serum ALT decreased more than 50% of the original value; Invalid: Failure to meet the above criteria

SECONDARY OUTCOMES:
The changes of ALT levels compared with baseline | less than 4 weeks
  ALT changes at other time points （1 week, 2 week, 3 week) compared with baseline
The changes of AST levels compared with baseline | less than 4 weeks
  AST changes at other time points （1 week, 2 week, 3 week) compared with baseline
The condition of acute liver injuries becomes the chronic liver disease | 6 months
  Proportion of patients with chronic drug-induced liver injury after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, M.D, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
Based on the principle of confidentiality of subjects' privacy and related information, this plan not to make IPD available to other researchers.

REFERENCES:
- [Background] Navarro VJ, Senior JR. Drug-related hepatotoxicity. N Engl J Med. 2006 Feb 16;354(7):731-9. doi: 10.1056/NEJMra052270. No abstract available. PMID 16481640
- [Background] Kullak-Ublick GA, Andrade RJ, Merz M, End P, Benesic A, Gerbes AL, Aithal GP. Drug-induced liver injury: recent advances in diagnosis and risk assessment. Gut. 2017 Jun;66(6):1154-1164. doi: 10.1136/gutjnl-2016-313369. Epub 2017 Mar 23. PMID 28341748
- [Background] Sgro C, Clinard F, Ouazir K, Chanay H, Allard C, Guilleminet C, Lenoir C, Lemoine A, Hillon P. Incidence of drug-induced hepatic injuries: a French population-based study. Hepatology. 2002 Aug;36(2):451-5. doi: 10.1053/jhep.2002.34857. PMID 12143055
- [Background] Bjornsson ES, Bergmann OM, Bjornsson HK, Kvaran RB, Olafsson S. Incidence, presentation, and outcomes in patients with drug-induced liver injury in the general population of Iceland. Gastroenterology. 2013 Jun;144(7):1419-25, 1425.e1-3; quiz e19-20. doi: 10.1053/j.gastro.2013.02.006. Epub 2013 Feb 16. PMID 23419359
- [Background] Vuppalanchi R, Liangpunsakul S, Chalasani N. Etiology of new-onset jaundice: how often is it caused by idiosyncratic drug-induced liver injury in the United States? Am J Gastroenterol. 2007 Mar;102(3):558-62; quiz 693. doi: 10.1111/j.1572-0241.2006.01019.x. PMID 17156142
- [Background] Wei G, Bergquist A, Broome U, Lindgren S, Wallerstedt S, Almer S, Sangfelt P, Danielsson A, Sandberg-Gertzen H, Loof L, Prytz H, Bjornsson E. Acute liver failure in Sweden: etiology and outcome. J Intern Med. 2007 Sep;262(3):393-401. doi: 10.1111/j.1365-2796.2007.01818.x. PMID 17697161
- [Background] Chalasani N, Bonkovsky HL, Fontana R, Lee W, Stolz A, Talwalkar J, Reddy KR, Watkins PB, Navarro V, Barnhart H, Gu J, Serrano J; United States Drug Induced Liver Injury Network. Features and Outcomes of 899 Patients With Drug-Induced Liver Injury: The DILIN Prospective Study. Gastroenterology. 2015 Jun;148(7):1340-52.e7. doi: 10.1053/j.gastro.2015.03.006. Epub 2015 Mar 6. PMID 25754159
- [Background] Danan G, Benichou C. Causality assessment of adverse reactions to drugs--I. A novel method based on the conclusions of international consensus meetings: application to drug-induced liver injuries. J Clin Epidemiol. 1993 Nov;46(11):1323-30. doi: 10.1016/0895-4356(93)90101-6. PMID 8229110
- [Background] Rockey DC, Seeff LB, Rochon J, Freston J, Chalasani N, Bonacini M, Fontana RJ, Hayashi PH; US Drug-Induced Liver Injury Network. Causality assessment in drug-induced liver injury using a structured expert opinion process: comparison to the Roussel-Uclaf causality assessment method. Hepatology. 2010 Jun;51(6):2117-26. doi: 10.1002/hep.23577. PMID 20512999
- [Background] Bjornsson ES, Hoofnagle JH. Categorization of drugs implicated in causing liver injury: Critical assessment based on published case reports. Hepatology. 2016 Feb;63(2):590-603. doi: 10.1002/hep.28323. Epub 2015 Dec 21. PMID 26517184
- [Background] Hoofnagle JH, Bjornsson ES. Drug-Induced Liver Injury - Types and Phenotypes. N Engl J Med. 2019 Jul 18;381(3):264-273. doi: 10.1056/NEJMra1816149. No abstract available. PMID 31314970
- [Background] Chen Y, Ye P, Ren C, Ren P, Ma Z, Zhang L, Zhou W, Jiang C. Pharmacoeconomics of three Therapeutic Schemes for Anti-tuberculosis Therapy Induced Liver Injury in China. Open Med (Wars). 2018 Mar 21;13:53-63. doi: 10.1515/med-2018-0010. eCollection 2018. PMID 29607414
- [Background] Naiqiong W, Liansheng W, Zhanying H, Yuanlin G, Chenggang Z, Ying G, Qian D, Dongchen L, Yanjun Z, Jianjun L. A Multicenter and Randomized Controlled Trial of Bicyclol in the Treatment of Statin-Induced Liver Injury. Med Sci Monit. 2017 Dec 4;23:5760-5766. doi: 10.12659/msm.904090. PMID 29200411
- See also: PMID: 28341748 — https://gut.bmj.com/content/66/6/1154
- See also: PMID: 23419359 — https://linkinghub.elsevier.com/retrieve/pii/S0016508513002175
- See also: PMID: 25754159 — https://linkinghub.elsevier.com/retrieve/pii/S001650851500311X
- See also: PMID: 8229110 — https://linkinghub.elsevier.com/retrieve/pii/0895435693901016
- See also: PMID: 29607414 — https://www.degruyter.com/document/doi/10.1515/med-2018-0010/html
- See also: PMID: 29200411 — https://medscimonit.com/abstract/index/idArt/904090